CLINICAL TRIAL: NCT07387770
Title: Assessment of Muscle Deterioration in Hospitalized Cancer Patients Using Surface Electromyography, Dynamometry, and Bioimpedance
Brief Title: Muscle Deterioration in Hospitalized Cancer Patient
Acronym: MUSONC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Inés Llamas-Ramos, Principal Investigator, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ONCO2026
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Oncologic Diseases
Keywords: cancer cachexia; sarcopenia; surface electromyography; bioimpedance analysis; hospitalized patients; protocol; muscle deterioration
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMG (Experimental): EMG screening
  Interventions: Diagnostic Test: Screenig Phase

INTERVENTIONS:
Diagnostic Test: Screenig Phase — EMG Parameters Analyzed:
  * Amplitude: Root mean square (RMS) during maximal voluntary contraction (MVC) and during sustained contraction, normalized to %MVC.
  * Frequency: Median frequency (MDF) and mean frequency (MNF) calculated using the fast Fourier transform (FFT) with 0.5-1 s sliding windows.
  Fatigue Indices
  * Rate of MDF decline (Hz/s) during sustained contraction.
  * Ratio of RMS at the end versus the beginning of the sustained contraction.
  * Time to task failure (s) during sustained effort.
  Quality Control:
  Quality control included real-time visual inspection of signals for movement artifacts, verification of baseline stability (resting activity <10-20 µV RMS), and complete post-acquisition review with exclusion of segments containing >20% artifact contamination.

SUMMARY:
Cancer cachexia and skeletal muscle deterioration represent significant challenges in oncology, affecting up to 42% of cancer patients and correlating with poor clinical outcomes, increased treatment toxicity, and reduced overall survival. Early identification of patients at risk through comprehensive musculoskeletal assessment is essential for timely therapeutic intervention.

This paper presents a detailed protocol for the longitudinal evaluation of skeletal muscle deterioration in hospitalized cancer patients using an integrated, multimodal approach. The protocol combines validated questionnaires (SARC-F, MSAS, EORTC QLQ-C30, and PSQI), functional measurements (handgrip strength), body composition analysis (bioelectrical impedance analysis), neuromuscular assessment (surface electromyography), and serum biomarkers (basic panel approach).

The study aims to recruit 45-50 patients with confirmed malignancy requiring hospitalization for ≥4 days, with daily functional measurements and biomarker evaluations at admission and discharge. The protocol prioritizes methodological rigor in vulnerable populations, incorporates standardized procedures for real-world clinical settings, and emphasizes quality control measures.

Expected outcomes include the identification of longitudinal patterns of muscle deterioration, validation of serum biomarker signatures for cachexia detection, and characterization of neuromuscular fatigue patterns using surface electromyography. This comprehensive framework addresses current gaps in skeletal muscle assessment during acute hospitalization and provides a foundation for future interventional studies. The protocol adheres to international ethical standards and considerations for research in vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 18 years
* Confirmed malignant neoplasm diagnosis
* Hospitalization anticipated for at least 4 days
* Capacity to provide informed consent and complete questionnaires
* ECOG performance status 0-3
* Ability to perform voluntary contractions of upper and lower extremities

Exclusion Criteria:

* Medical contraindications to strength testing (recent fractures, acute injuries) - Severe neurological impairment precluding functional assessment
* Implanted electronic devices (relative contraindication for bioimpedance)
* Severe cognitive impairment preventing questionnaire completion
* Extensive skin lesions preventing electrode placement for sEMG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SARC-F Sarcopenia Screening Tool | Baseline and up to 10 days
  The SARC-F questionnaire (Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls) will be administered to all participants at baseline and at discharge. This five-item instrument evaluates functional limitations, with total scores ranging from 0 to 10; scores ≥4 indicate an increased risk of sarcopenia. The SARC-F demonstrates a sensitivity of 71-89% and a specificity of 84-91% for sarcopenia detection across diverse populations.
Symptoms prevalence. Memorial Symptom Assessment Scale (MSAS) | Baseline and and up to 10 days
  The Memorial Symptom Assessment Scale (MSAS) will be administered using the validated Spanish version by Llamas-Ramos et al. The 24-item short form (MSAS-SF) assesses symptom frequency, severity, and associated distress across three core dimensions: the Global Distress Index, the Physical Symptom Subscale, and the Psychological Symptom Subscale. The instrument has demonstrated excellent psychometric properties in Spanish-speaking cancer populations (Cronbach's α > 0.80) and superior sensitivity to symptom changes compared with single-item scales.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Baseline and and up to 10 days
  The EORTC QLQ-C30 is the gold-standard instrument for assessing quality of life in cancer patients. This 30-item questionnaire evaluates five functional scales (physical, role, emotional, cognitive, and social functioning), global health status/quality of life, symptom scales (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, and diarrhea), and financial difficulties. Scores are linearly transformed to 0-100 scales, with higher scores indicating better functioning on functional scales and greater symptom burden on symptom scales. The EORTC QLQ-C30 has demonstrated prognostic validity for survival outcomes across multiple cancer types.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and up to 10 days
  The Pittsburgh Sleep Quality Index (PSQI) evaluates sleep quality over the preceding month using 19 self-reported items, yielding seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). The global PSQI score ranges from 0 to 21, with scores >5 indicating poor sleep quality. Among cancer patients, the PSQI demonstrates 89.6% sensitivity and adequate psychometric properties for detecting sleep disturbances.
Bioimpedance Electrical Analysis | Baseline and and up to 10 days
  Bioelectrical Impedance Analysis (BIA) will be performed using InBody equipment (bipedal configuration, 50 kHz impedance measurement). Standardized protocols will include: (1) 4-6 h of fasting, when feasible; (2) micturition 30 min prior to assessment; (3) a 15-min supine rest period to allow for fluid redistribution; and (4) documentation of hydration status using a structured clinical scale.
Handgrip Strength Assessment | Baseline and through study completion, an average of 10 days
  Handgrip strength will be measured daily using a calibrated digital dynamometer (EH101, China), following the American Society of Hand Therapists (ASHT) protocol. Prior to study initiation, the dynamometer underwent precision testing using calibrated weights (error <5%) and reliability assessment in 12 healthy volunteers (ICC = 0.92, 95% CI: 0.86-0.96).
Surface Electromyography Assessment | Baseline and through study completion, an average of 10 days
  Surface electromyography (sEMG) will be acquired using the mDurance system (Shimmer3 wireless hardware), with a sampling rate of 1000 Hz, band-pass filtering from 10 to 500 Hz, and a 50 Hz notch filter to eliminate power-line interference.
  Electrode Preparation and Placement Skin will be prepared by shaving with disposable razors, gentle abrasion with fine-grit sandpaper, and cleansing with 70% alcohol, followed by complete air-drying. Disposable Ag/AgCl electrodes (20 mm interelectrode distance, in accordance with SENIAM recommendations) will be placed using precise anatomical landmarks on the vastus lateralis, vastus medialis, and upper trapezius muscles.

SECONDARY OUTCOMES:
Blood sample collection | Baseline and up to 10 days
  Blood samples will be collected during routine morning laboratory draws at admission and discharge, with additional volumes (10-15 mL) obtained for research purposes. Serum will be separated via centrifugation at 3000 rpm for 10 minutes and stored at -80°C until batch analysis. All analytical procedures will be performed in accordance with standard hospital clinical laboratory protocols.

IPD SHARING:
Plan to Share IPD: No